CLINICAL TRIAL: NCT05206539
Title: Efficacy of Self-assembling Peptide P11-4, Casein Phosphopeptide - Amorphous Calcium Fluoride Phosphate and Resin Infiltrant in Treatment of Initial Caries on Smooth Surfaces in Permanent Teeth in Children
Brief Title: Efficacy of Different Agents in Treatment of Initial Caries on Smooth Surfaces in Permanent Teeth in Children
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Plovdiv Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: MU_WSL
Record Dates: First submitted 2022-01-12; First posted 2022-01-25 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-02

CONDITIONS: White Spot Lesion of Tooth
Keywords: white spot lesions; initial caries; early caries lesions; self-assembling peptide p11-4; cpp-acfp; resin infiltrant; icon infiltration; non-operative dental treatment
MeSH Terms: interventions — casein phosphopeptide-amorphous calcium phosphate nanocomplex; Control Groups

STUDY DESIGN:
Intervention Model Description: The trial to be conducted is a randomized controlled clinical crossover experimental study with split-mouth design. The within-subject design randomly allocates experimental and control interventions to different areas in the oral cavity (teeth, surfaces, arches, quadrants) and has the advantage of reducing outcome variability estimation since each patient is its own control, leading to potential increase in statistical power.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: This is a double-blinded trial, i.e., where patients and outcomes assessor are not aware which white spot lesion what treatment will receive, unlike the operator which is not blinded for the study due to the nature of the investigated techniques.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SAP11-4 group (Gr CR) (Experimental): The Gr CR will receive treatment with Curodont RepairTM (Credentis; Windisch, Switzerland), according to the manufacturer's instructions.
  Interventions: Drug: Self-assembling peptide (P11-4)
- CPP-ACFP group (Gr V) (Active Comparator): The Gr V will receive treatment with MI varnishTM (GC Corporation, Tokyo, Japan), according to the manufacturer's instructions.
  Interventions: Drug: CPP-ACFP
- Resin infiltration group (Gr I) (Active Comparator): The Gr I receive treatment with Icon Vestibular (DMG, Germany), according to the manufacturer's instructions.
  Interventions: Drug: Resin infiltration
- Control group (Gr NT) (Placebo Comparator): The control group (Gr NT) receive no intervention except brushing twice daily with aminofluoride toothpaste and toothbrush provided by researcher.
  Interventions: Other: Control Group, No Treatment

INTERVENTIONS:
Drug: Self-assembling peptide (P11-4) — Prior to application, teeth are isolated by cotton rolls and gently air dried. The surface of the lesion is conditioned with a 2% sodium hypochlorite solution for 20 s and then rinse with water. Application of 35% phosphoric acid etching gel for 20 sec followed by rinsing with water-air spray for 30 sec. Drying the surface with compressed oil-free air for 60 sec. Curodont Repair is dissolve in 0.05 ml of distilled water and applied to the surface and allowed to work for about 5 min.
  Participants will receive oral hygiene instructions.
  Other Names: Curodont Repair
  Arms: SAP11-4 group (Gr CR)
Drug: CPP-ACFP — Prior to application, teeth are isolated by cotton rolls and gently air dried. Application of fluoride varnish with a brush applicator on the surface of the teeth for 5 minutes. Patients is advising not to brush their teeth or chew food for at least 4 h after treatment.
  Participants will receive oral hygiene instructions
  Other Names: MI varnishTM (GC Corporation, Tokyo, Japan); RecaldentTM (CPP-ACP)
  Arms: CPP-ACFP group (Gr V)
Drug: Resin infiltration — The validated ICON Vestibular (DMG) infiltration lesion infiltration protocol is applied. Icon Etch (DMG) etching gel containing 15% hydrochloric acid is applied for 120 seconds using an applicator. It is then removed by rinsing thoroughly with water-air spray for 30 seconds. Then follows application of pure alcohol - Icon Dry (DMG) for 30 seconds for complete drying of the lesion and additional drying compressed oil-free air for 40 sec. Application of Icon Infiltrant (DMG) using a microapplicator allows it to penetrate for 3 minutes, during which, if necessary, it is reapplied several times. Excess material is removed with dry microbrushes and followed by light curing for 40 seconds. Re-applying of the infiltrate for 1 minute, removal of excess material, light curing for 40 seconds. Participants will receive oral hygiene instructions
  Other Names: Icon Vestibular (DMG; Hamburg, Germany)
  Arms: Resin infiltration group (Gr I)
Other: Control Group, No Treatment — Everyday oral hygiene instructions Subjects will receive non-prescription fluoride toothpaste (1400 ppm Fluoride, Elmex junior) and oral hygiene instructions. The dosage will be 1/2 inch strip of paste 2x/day for 8 weeks. Subjects will apply paste to a toothbrush and brush teeth thoroughly for at least 1 minute then expectorate and rinse.
  Other Names: Home Oral Care
  Arms: Control group (Gr NT)

SUMMARY:
White spot lesions (WSL) are characterized by an apparently intact outer surface and a demineralized subsurface, and are considered the first clinical sign of dental caries.

Aim of this study is to determine the treatment potential of self-assembling peptide (P11-4), casein phosphopeptide-amorphos calcium fluoride phosphate (CPP-ACFP) and resin infiltration technique to reverse or arrest the WSLs in the same oral environments in pediatric patients using visual assessments and laser fluorescence investigation.

DETAILED DESCRIPTION:
White spot lesions (WSL) are characterized by an apparently intact outer surface and a demineralized subsurface, and are considered the first clinical sign of dental caries. These lesions are characterized by white chalky appearance. As caries is reversible under favorable conditions, many approaches have focused on treating it as soon as possible1.

Aim of this study is to determine the treatment potential of self-assembling peptide (P11-4), casein phosphopeptide-amorphos calcium fluoride phosphate (CPP-ACFP) and resin infiltration technique to reverse or arrest the WSLs in the same oral environments in pediatric patients. This will be achieved using visual assessments and laser fluorescence investigation.

The proposed study is a randomized controlled clinical trial with split-mouth design. Included are forty positive patients aged 9-17 years, with at least four visible WSL on smooth surfaces in permanent teeth, requiring non-operative treatment. WSL will be assessed visually by ICDAS II, Nyvad criteria and laser fluorescence (LF pen). The lesions are randomly assigned into 4 groups (n = 40): Gr NT (no treatment, control group), Gr CR (Curodont Repair), Gr V (MI Varnish), Gr I (Icon) groups. Lesions will be assessed by International Caries Detection and Assessment System, Nyvad caries activity criteria and laser fluorescence at baseline and follow-up period after1, 3, 6 and 12 months.

Data will be analyzed with intention-to-treat concept by Student T-test for paired samples, Wilcoxon signed rank test, P< .05. Pre-test on 20 subjects resulted in n=41 patients sample size.

ELIGIBILITY:
Inclusion Criteria:

* Participants in the study are children 9 to 17 years old.
* Obtained written informed consent from parents or gave-givers as well as obtained verbal informed consent from the child to participate in the study, in which procedures are explained in age-appropriate manner.
* Children, identified as positive or definitely positive through Frankl behavioral rating scale.
* Presence of at least four initial carious lesions of smooth surface (white spots) in permanent teeth that reach the inside of the enamel but are not cavitated, estimated with ICDAS system values 01 (first visible enamel change) and 02 (localized visible enamel change), Nyvad caries activity criteria (1 -active, noncavited lesion) and DIAGNOdent pen values up to 24.
* Study participants did not conduct remineralizing or topical fluorine therapy of the lesions involved up to six months prior to inclusion in the study.
* Children without a history of allergy to the administered medications

Exclusion Criteria:

* Patients with general diseases or conditions associated with decreased salivation and intake of medications suppressing salivary current. Children with cognitive and behavioral disorders. The presence of a disease is confirmed by an anamnestic interview with the parent.
* Children with a history of allergy to the administered medications
* Patient with non-carious lesion such as enamel hypoplasia, or any developmental defects.
* Patient received restorations or any remineralizing agent other than the regular toothpaste during the last 6 months.
* Participant in another trial.

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Change in lesion fluorescence evaluated using diode laser fluorescence device. | 12 months: (Baseline, 1 month, 3 months, 6months and 12 months)
  Laser fluorescence values are categorized: 20-24
  * Category 0= LF values 0-7, caries-free enamel surface
  * Category 1=LF values 8-14, caries extending up to halfway through the enamel
  * Category 2=LF values 15-24, caries in the inner half of enamel
  * Category 3= LF values >24, caries in dentine

SECONDARY OUTCOMES:
Visual assessment using ICDAS II coding system | 12 months: (Baseline, 1 month, 3 months, 6months and 12 months)
  Code 0 Sound tooth surface:
  Code 1: First visual change in enamel. Code 2: Distinct visual change in enamel visible when wet, lesion must be visible when dry.
  Code 3: Localized enamel breakdown because of caries with no visible dentin or underlying shadow.
  Code 4: Underlying dark shadow from dentin with or without localized enamel breakdown.
  Code 5: Distinct cavity with visible dentin. Code 6: Extensive distinct cavity with visible dentin. After treatment, the evaluation will be performed as follows. If the score has increased to ICDAS 3 or more indicates caries progression and if it decreases to 0-1 this indicates caries regression; if score remains the same this indicates no change in lesion. No. of lesions with scores 0,1,2,3 or more will be assessed and analyzed.
Activity of a carious lesion using Nyvad Caries Diagnostic Criteria | 12 months: (Baseline, 1 month, 3 months, 6months and 12 months)
  Code 0: Sound - Normal enamel Code 1: Active caries (intact surface) - Surface of enamel is whitish/yellowish opaque Code 2: Active caries (surface discontinuity) Code 3: Active caries (cavity) - Enamel/dentin cavity easily visible with the naked eye.
  Code 4: Inactive caries (intact surface) - Surface of enamel is whitish, brownish or black.
  Code 5: Inactive caries (surface discontinuity) - Same criteria as score 4. Localized surface defect (microcavity) in enamel only Code 6: Inactive caries (cavity) - Enamel/dentin cavity easily visible with the naked eye; surface of cavity may be shiny and feels hard on probing with gentle pressure.
  Code 7: Filling (sound surface) Code 8: Filling + active caries - Caries lesion may be cavitated or noncavitated.
  Code 9: Filling + inactive caries - Caries lesion may be cavitated or noncavitated.

CONTACTS AND LOCATIONS:
Overall Officials: Ani Belcheva, PhD, Study Director — Medical University Plovdiv, Bulgaria
Locations (1):
- Department of Pediatric Dentistry, Faculty of Dental Medicine, Medical University - Plovdiv, Plovdiv, Bulgaria

IPD SHARING:
Plan to Share IPD: No